CLINICAL TRIAL: NCT04931095
Title: The Impact of Oral Cannabis Administration and Co-Administration of Alcohol on Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00290015; 1R01DA052295-01 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Cannabis Intoxication; Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — nabiximols; Ethanol

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind (Participant, Outcomes Assessor), placebo controlled, and double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo cannabis + placebo alcohol (Placebo Comparator): Participants administer oral cannabis containing 0mg THC in combination with a placebo alcohol drink.
  Interventions: Drug: Cannabis; Drug: Alcohol
- low dose cannabis with placebo alcohol (Experimental): Participants administer oral cannabis containing 10mg THC in combination with a placebo alcohol drink.
  Interventions: Drug: Cannabis; Drug: Alcohol
- high dose cannabis with placebo alcohol (Experimental): Participants administer oral cannabis containing 25mg THC in combination with a placebo alcohol drink.
  Interventions: Drug: Cannabis; Drug: Alcohol
- low dose cannabis with low dose alcohol (Experimental): Participants administer oral cannabis containing 10mg THC in combination with an alcohol drink (0.05 percent BAC).
  Interventions: Drug: Cannabis; Drug: Alcohol
- high dose cannabis with low dose alcohol (Experimental): Participants administer oral cannabis containing 25mg THC in combination with an alcohol drink (0.05 percent BAC).
  Interventions: Drug: Cannabis; Drug: Alcohol
- Placebo cannabis + low dose alcohol (Experimental): Participants administer oral cannabis containing 0mg THC in combination with an alcohol drink (0.05 percent BAC).
  Interventions: Drug: Cannabis; Drug: Alcohol
- Placebo cannabis + high dose alcohol (Experimental): Participants administer oral cannabis containing 0mg THC in combination with an alcohol drink (0.08 percent BAC).
  Interventions: Drug: Cannabis; Drug: Alcohol

INTERVENTIONS:
Drug: Cannabis — Cannabis will be orally ingested via a brownie
Drug: Alcohol — Alcohol will be orally ingested via a flavored drink

SUMMARY:
This study will evaluate the individual and interactive effects of oral cannabis and alcohol on subjective and behavioral measures of impairment.

DETAILED DESCRIPTION:
This clinical laboratory study will be double-blind, placebo-controlled and will utilize a within-subjects experimental design. Participants will complete 7 outpatient drug administration sessions that will consist of self-administration of oral cannabis (0, 10 or 25mg THC) and alcohol (either placebo or active; BAC of 0.05 percent); participants will always receive both an alcohol drink (active or placebo) and dose of cannabis (active or placebo). Participants will also complete a condition in which they administer alcohol (BAC: 0.08 percent) with placebo cannabis, as a positive control. Primary outcomes include performance on field sobriety tests, cognitive and psychomotor impairment, subjective drug effects, and simulated driving performance. Blood concentrations of THC and THC metabolites will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 21 and 55
3. Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
4. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at each study visit.
5. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
6. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
7. Have not donated blood in the prior 30 days.
8. Report at least 2 days of binge drinking in the past 90 days (greater than 4 or 5 drinks on a single occasion for women and men, respectively)
9. Report ≥ 1 use of cannabis in the past year
10. Provide negative urine test for illicit drug use (excluding THC) and negative breath alcohol test (0% BAC) at screening and before study sessions
11. Report at least 1 instance of simultaneous alcohol and use in the past year.

Exclusion Criteria:

1. Psychoactive drug use (aside from cannabis, nicotine, alcohol, or caffeine) in past month
2. Current use of over-the-counter (OTC) drugs, supplements/vitamins, or prescription medications that, in the opinion of the investigator or medical staff, will impact the participant's safety
3. History of or current evidence of significant medical condition
4. Evidence of current psychiatric condition [(MINI for Diagnostic and Statistical Manual (DSM)-V)]
5. Meet criteria for severe alcohol use disorder (MINI for DSM-V)
6. Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-Ar) score > 9
7. Been in treatment previously for alcohol or cannabis use disorder
8. Use of cannabis, on average, more than 2 times/week over past 3 months
9. Liver function tests more than 2x normal range
10. Enrollment in another clinical trial or receiving of any drug as part of research within past 30 days
11. Shipley vocabulary score <18 (corresponds to 5th grade reading level).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
DRUID application global impairment score | 7.5 hours
  Acute cognitive and behavioral impairment will be assessed with global impairment score(range 0-100) on the DRUID app (higher scores indicate greater impairment).
Correct Trials on Paced Auditory Serial Addition Task (PASAT) | 7.5 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Will report the total correct trials out of 90 recorded (lower scores indicate worse performance).
Correct Trials on the Digit Symbol Substitution Task (DSST) | 7.5 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Will report the total correct trials in 90 seconds (lower scores indicate worse performance).
Cumulative score on Field Sobriety Tests | 7.5 hours
  Impairment will be assessed using a battery of standard field sobriety tests including: the Horizontal Gaze Nystagmus Test (HGN), the Walk and Turn, the One Leg Stand, and the Modified Romberg Balance. We will report the cumulative amount of clues observed across these tasks (out of a possible 22 clues).
Drug Effect Questionnaire (DEQ) - Feel Drug Effect | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "feel drug effects". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Feel High | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "feel high". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Confidence to Drive | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "confidence to drive". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Willingness to Drive | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "willingness to drive". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Biphasic alcohol effects scale (BAES) - Sedative Score | 7.5 hours
  The BAES is used to assess sedative and stimulant subjective effects of alcohol. There are 7 sedative-related questionnaire items, each presented on a scale of 0 (not at all) to 10 (extremely), which are integrated to produce an overall sedative score (0-70).
Biphasic alcohol effects scale (BAES) - Stimulant Score | 7.5 hours
  The BAES is used to assess sedative and stimulant subjective effects of alcohol. There are 7 stimulant-related questionnaire items, each presented on a scale of 0 (not at all) to 10 (extremely), which are integrated to produce an overall stimulant score (0-70).
Subjective high assessment scale (SHAS) | 7.5 hours
  For the SHAS, participants are presented with 13 questionnaire items, displayed on a visual analog scale anchored from 0 (normal) to 10 (extremely), which assess subjective effects of alcohol. These items are integrated to produce an overall SHAS score (0-130)
Driving performance as assessed by standard deviation of lateral position (SDLP) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. SDLP (measured in cm) will be determined during each drive. This measure is a composite index of lateral control and incorporates lane weaving, swerving, and over-correcting. SDLP is the gold standard of quantifying the magnitude of driving impairment from drugs and alcohol and has excellent predictive validity to actual driving. Scores range from 0 to no upper limit. Higher scores represent higher magnitude of driving impairment.
Driving performance as assessed by composite drive score | 7.5 hours
  Driving impairment will be assessed via a composite drive score (higher scores indicate greater impairment). The composite drive score is derived by integrating various driving outcomes (see primary and secondary driving outcomes). There is no upper or lower limit to possible scores

SECONDARY OUTCOMES:
Driving performance as assessed by standard deviation of speed (SDSP) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. SDSP will be determined during each drive; this measure quantifies the variability in speed (in MPH) observed.
Driving performance (mean speed) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. Mean speed (in MPH) over the course of each drive will be determined.
Driving performance (number of speed exceedances) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The cumulative number of times participants exceed the allowable speed limit during each drive.
Driving performance (number of accidents) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The cumulative number of accidents (including car collisions, pedestrians hit, etc.) during each drive.
Driving performance (total rule violations) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The cumulative number of rule violations (including number of missed stop signs, illegal turns, speed exceedances, etc.) during each drive.
Driving performance (distance to lead vehicles) | 7.5 hours
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. The mean distance (in meters) maintained to lead vehicles during car-following segments of each drive.
Attempted Trials on the Digit Symbol Substitution Task (DSST) | 7.5 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. The number of attempted trials will be recorded
Percentage Correct on attempted trials on the Digit Symbol Substitution Task (DSST) | 7.5 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Percentage of correct trials out of those attempted will be recorded
Reaction time on Paced Auditory Serial Addition Task | 7.5 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. The mean reaction time (in milliseconds) to select correct responses will be recorded.
Field Sobriety Test - Score on Horizontal Gaze Nystagmus Test | Up to 7.5 hours
  Impairment will be assessed using performance on the Horizontal Gaze Nystagmus Test (HGN). Total score will be recorded (out of possible 6 clues) with higher scores indicating higher impairment.
Field Sobriety Test - Score on Walk and Turn test | Up to 7.5 hours
  Impairment will be assessed using performance on the the Walk and Turn. Total score will be recorded (out of a possible 8 clues) with higher scores indicating higher impairment.
Field Sobriety Test - Score on One Leg Stand | Up to 7.5 hours
  Impairment will be assessed using performance on the One Leg Stand test. Total score will be recorded (out of a possible 4 clues) with higher scores indicating higher impairment.
Field Sobriety Test - Score on Modified Romberg Balance | Up to 7.5 hours
  Impairment will be assessed using performance on the Modified Romberg Balance test. Total score will be recorded (out of a possible 4 clues) with higher scores indicating higher impairment.
Drug Effect Questionnaire - Like Drug Effect | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "like drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Want more | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "want more". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Dislike Drug Effect | 7.5 hours
  The DEQ will be used to obtain subjective ratings of "dislike drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Pharmacokinetics - CMax for THC and THC metabolites | 7.5 hours
  Whole blood concentrations of THC, 11-OH- THC, and THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentration (Cmax) is determined as the highest concentration reached for each individual. Characterizing these cannabinoids will allow for adequate control for individual differences in drug absorption and metabolism in statistical analyses and assist with interpretation of subjective and behavioral outcomes.
Pharmacokinetics - AUC for THC and THC metabolites | Up to 7.5 hours
  Whole blood concentrations of THC, 11-OH- THC, and THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline. Characterizing these cannabinoids will allow for adequate control for individual differences in drug absorption and metabolism in statistical analyses and assist with interpretation of subjective and behavioral outcomes.
Pharmacokinetics - Breath Alcohol Concentration (BAC) | Up to 7.5 hours
  BAC will be measured using the Alco-Sensor IV. Measuring BAC is needed to confirm that participants reached the targeted BAC for a given session and to confirm adherence to pre-session alcohol abstinence requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No